CLINICAL TRIAL: NCT01893216
Title: Study of Possible Interactions Between Psychiatric Disorders and Sexual Dysfunction in Infertile Men
Brief Title: Risk Factors of Psychiatric Disorders and Sexual Dysfunction in Infertile Men
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Wan Zi, Doctor, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: IMPsySex
Record Dates: First submitted 2013-07-02; First posted 2013-07-08 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Anxiety; Depression; Sexual Dysfunction; Infertility
Keywords: anxiety; depression; sexual dysfunction; infertility
MeSH Terms: conditions — Anxiety Disorders; Depression; Sexual Dysfunction, Physiological; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- with depression or anxiety: Hospital Anxiety and Depression Scale score over 9 points
- without depression or anxiety: Hospital Anxiety and Depression Scale score less than 8 points

SUMMARY:
To investigate the prevalence of psychological symptoms and sexual dysfunction, and to estimate their possible interactions in infertile men.

DETAILED DESCRIPTION:
Although psychological disorders such as anxiety and depression are known to be associated with sexual dysfunction, and their interactions have been reported by many studies, particularly the prevalence of these two aspects and the relationship between them in infertile men in China have not been well investigated.

The investigators' aim is to evaluate the prevalence of psychological symptoms and sexual dysfunction and interactions between them systematically by using validated questionnaires and scales.

ELIGIBILITY:
Inclusion Criteria:

* men who seek treatment for infertility (infertility is defined as the inability to conceive after 1 year of unprotected intercourse)
* age ≥ 18 years
* in a heterosexual, stable relationship for at least 1 year
* able to read and speak Chinese

Exclusion Criteria:

* inability to read and understand the questionnaire because of language difficulties
* already evaluated during an earlier survey
* men on medication that could have affected their ejaculatory and erectile function and/or psychological status

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: male outpatients visiting the Centre of Reproduction at First Affiliated Hospital of Sun Yat-sen University
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-08 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Incidence and Risk Factors of sexual dysfunction and psychological disorders in infertile men | one year

SECONDARY OUTCOMES:
Interactions between Psychiatric Disorders and Sexual Dysfunction in Infertile Men | one year

CONTACTS AND LOCATIONS:
Overall Officials: Chunhua Deng, MD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China